CLINICAL TRIAL: NCT02208388
Title: Prospective Evaluation of MyocaRdial PerFUSion ComputEd Tomography Trial: Ischemia-guided Revascularization Using Perfusion Coronary CT vs. Fractional Flow Reserve
Brief Title: Prospective Evaluation of MyocaRdial PerFUSion ComputEd Tomography Trial
Acronym: PERFUSERCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Young-Hak Kim, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Young-Hak Kim, MD, PhD, MD, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMCCV2014-06
Record Dates: First submitted 2014-07-31; First posted 2014-08-05 (Estimated); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Coronary Disease
Keywords: Computed tomography perfusion; Fractional flow reserve
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computed tomography perfusion (Experimental): Patients with Computed tomography perfusion
  Interventions: Device: computed tomography perfusion guided treatment
- Fractional flow reserve (Active Comparator): Patients with Fractional flow reserve
  Interventions: Device: Fractional flow reserve guided treatment

INTERVENTIONS:
Device: computed tomography perfusion guided treatment
  Arms: Computed tomography perfusion
Device: Fractional flow reserve guided treatment
  Arms: Fractional flow reserve

SUMMARY:
The purpose of this study is to evaluate safety and effectiveness of CTP(computed tomography perfusion) guided revascularization vs FFR(Fractional flow reserve) guided revascularization

ELIGIBILITY:
Inclusion Criteria:

* Age 20 and more
* Diagnosed angina or angina equivalent symptom or positive exercise treadmill test
* Patients with intermediate- or high-risk probability of CAD defined by Diamond and Forester
* 70 % stenosis or more in coronary CTA
* Willing to provide informed, written consent

Exclusion Criteria:

* Requirement for surgical procedure
* Cardiogenic shock and/or need for mechanical/pharmacologic hemodynamic support
* Recent STEMI (<5 days)
* Non STEMI, if the cardiac troponin is not stable or starting to decline
* Left ventricular ejection fraction <30%
* Life expectancy <2 years
* Impaired renal function with an effective glomerular filtration rate less than 30mL/min/1.73 ㎡ or creatinine more than 2.0 mg/dL
* Undergoing evaluation for organ transplantation
* Participation or planned participation in another cardiovascular clinical trial
* Pregnancy
* Inability to take dual antiplatelet therapy for six months
* Previous CABG
* Left main disease requiring revascularization
* Any target lesion with in-stent restenosis
* NYHA class 3 or 4a
* Severe and persistent angina with severe limitation in everyday living activities (Canadian Cardiovascular Society grading Class IV)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2014-08-12 (Actual); Primary Completion 2028-03-05 (Estimated); Study Completion 2028-03-05 (Estimated)

PRIMARY OUTCOMES:
Composite Events | 1 year
  All cause death, Myocardial infarction, Diseased-related unplanned hospitalization or stroke

SECONDARY OUTCOMES:
All cause death | 5 year
  All cause death
Myocardial infarction | 5 year
  Myocardial infarction
Target vessel revascularization | 5 year
  Target vessel revascularization
Stent thrombosis | 5 year
  Stent thrombosis
Seattle Angina Questionnaire,EQ5D questionnaire | 5 year
  Quality of life score assessed by the EQ-5D-5L The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
  Higher score of EQ-5D and EQ VAS means the low quality of life. EQ-5D: the minimum and maximum values are 5 and 25 respectively. EQ VAS: the minimum and maximum values are 0 and 100 respectively.
  Seattle Angina Questionnaire The Seattle Angina Questionnaire (SAQ) is a vali- dated disease-specific instrument for assessing the health status of patients with coronary artery disease.
  SAQ scores can be aligned with clinical constructs (eg, scores on the SAQ angina frequency scale of 0-30 points indicate daily angina, 31-60 points indicate weekly angina, 61-99 points indicate monthly angina, and 100 points indicate no angina)
Success of intervention | 5 year
  Defined as mean lesion diameter stenosis ≤50% and without the occurrence of in-hospital myocardial infarction (MI), target vessel revascularization (TVR), or death
Cost effective analysis | 1 year
  Cost effective analysis

CONTACTS AND LOCATIONS:
Overall Officials: Byoung-Wook Choi, MD, Principal Investigator — Severance Hospital, Yonsei University College of Medicine; Young-Hak Kim, MD, Principal Investigator — Asan Medical Center
Locations (7):
- South Korea (7):
  - Asan Medical Center, Seoul, Songpa-Gu
  - Hallym University Sacred Heart Hospital, Anyang
  - Gangwon National Univ. Hospital, Chuncheon
  - Keimyung University Dongsan Medical Center, Daegu
  - Pusan National University Hospital, Pusan
  - Pusan National University Yangsan Hospital, Pusan
  - Severance Hospital, Seoul